CLINICAL TRIAL: NCT02977754
Title: Exploring the Prognostic Role of 18F-FDG PET/CT Imaging in Patients Affected by Hepatocellular Carcinoma (HCC) and Candidate to Treatment With Sorafenib
Brief Title: 18F-FDG PET in HCC Patients Candidate to Treatment With Sorafenib
Status: Completed | Type: Observational
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Other Study IDs: 1458
Record Dates: First submitted 2016-11-18; First posted 2016-11-30 (Estimated); Last update posted 2020-10-01 (Actual); Status verified 2020-09

CONDITIONS: HCC

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: This is an observational study — Imaging

SUMMARY:
The principal objective of this study is to explore the role of 18F-FDG PET in identifying sorafenib-induced metabolic shift in HCC, thus in predicting treatment response and disease outcome in advanced HCC patients candidate to systemic treatment with sorafenib.

DETAILED DESCRIPTION:
Aerobic glycolysis also called "Warburg effect", represents one of the distinctive hallmarks of the malignant cells. Although energetically less efficient than respiration, fermentative metabolism is advantageous for cell growth due to the increased availability of anabolic intermediates and the reduced cell dependence on oxygen. Moreover, by increasing intracellular reducing equivalents and decreasing mitochondria-derived ROS, glycolysis protects malignant cells from oxidant-induced senescence and apoptosis.

In diagnostic imaging, the "Warburg effect" is visualized thanks to the utilization of ﬂuoro-2-deoxyglucose, a glucose analogue, labeled with the positron emitting nuclide fluoride-18 (18F). F-2-ﬂuoro-2-deoxyglucose (18F-FDG) with positron emission tomography (PET) has emerged useful in many tumor types and in HCC can help ruling out extra-hepatic metastases or sites of recurrent disease, and giving prognostic information. Considering the abovementioned premises, the investigators hypothesize a potential use of 18F-FDG PET for the early assessment of sorafenib-induced metabolic shift in HCC, especially in well-differentiated subtypes usually showing an uptake of the tracer not different or at least not sufficiently increased compared to the normal liver.

For these reasons the investigators decided to conduct an explorative study for the assessment of predictive and prognostic role of 18F-FDG PET in patients affected by advanced HCC and candidate to systemic treatment with sorafenib.

The principal objective of this study is to explore the role of 18F-FDG PET in identifying sorafenib-induced metabolic shift in HCC, thus in predicting treatment response and disease outcome in advanced HCC patients candidate to systemic treatment with sorafenib.

More specifically the investigators will:

* compare 18F-FDG uptake in HCC lesions, identified as target lesions (diam. min. 2cm), at baseline, at 24 hours and 1 week after the first administration of sorafenib.
* correlate the patterns of 18F-FDG uptake in HCC lesions with objective tumor response assessed 8 weeks after the first administration of sorafenib according to mRECIST criteria.
* correlate the patterns of 18F-FDG uptake in HCC lesions with alpha-fetoprotein (AFP) variation at baseline, at 24 hours and 1 week after the first administration of sorafenib.
* correlate the patterns of 18F-FDG uptake in HCC lesions with progression-free survival (PFS) and overall survival (OS).

ELIGIBILITY:
Inclusion Criteria:

* patients with an histological diagnosis of HCC and scheduled to undergo systemic treatment with sorafenib;
* obtained informed consent

Exclusion Criteria:

* patients age <18 years
* pregnancy or breast-feeding;
* patients affected by other malignancies within the last 3 years, with the exception of surgically cured carcinoma in situ of the cervix, in situ breast cancer, incidental finding of stage T1a or T1b prostate cancer, and basal/squamous cell carcinoma of the skin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a single-center, single-arm study, lasting 36 months including an estimated period of 24 months for the enrolment and max 12 months of follow-up. All patients affected by HCC and referred to our Institution for systemic treatment with sorafenib will be evaluated for enrolment. A minimum number of 10 patients will be considered for the analysis.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2016-01; Primary Completion 2018-12 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Early change of metabolic characteristics (i.e. SUVmax, SUVmean, MTV, TLG) of HCC lesions under Sorafenib | Compare 18F-FDG uptake in HCC lesions at baseline and at 24 hours after the first administration of sorafenib.
  Baseline parameters

SECONDARY OUTCOMES:
Change of metabolic characteristics (i.e. SUVmax, SUVmean, MTV, TLG) of HCC lesions under Sorafenib | Compare 18F-FDG uptake in HCC lesions at baseline and 1 week after the first administration of sorafenib.
  Variation of parameters
Predictive role of metabolic characteristics of HCC (i.e. SUVmax, SUVmean, MTV, TLG) lesions under Sorafenib | Correlate the patterns of 18F-FDG uptake in HCC lesions with objective tumor response assessed 8 weeks after the first administration of sorafenib according to mRECIST criteria
  PET scan parameters compared to response
Prognostic role of metabolic characteristics (i.e. SUVmax, SUVmean, MTV, TLG) of HCC lesions under Sorafenib | Correlate the patterns of 18F-FDG uptake in HCC lesions with progression-free survival (PFS) and overall survival (OS) assessed during a minimun of 12 months of follow up
  PET scan parameters compared to outcome

OTHER OUTCOMES:
Correlate tumor markers with metabolic characteristics (i.e. SUVmax, SUVmean, MTV, TLG) of HCC lesions under Sorafenib | Correlate the patterns of 18F-FDG uptake in HCC lesions with alpha-fetoprotein (AFP) measured at baseline and after 8 weeks of treatment
  PET scan parameters compared to tumor markers

CONTACTS AND LOCATIONS:
Overall Officials: Egesta Lopci, Principal Investigator — Istituto Clinico Humanitas
Locations (1):
- Istituto Clinico Humanitas, Rozzano, Milano, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Castello A, Rimassa L, Personeni N, Pressiani T, Smiroldo V, Lopci E. Metabolic Switch in Hepatocellular Carcinoma Patients Treated with Sorafenib: a Proof-of-Concept Trial. Mol Imaging Biol. 2020 Oct;22(5):1446-1454. doi: 10.1007/s11307-020-01489-6. PMID 32206991